CLINICAL TRIAL: NCT03778710
Title: Effect of Lymph Node Ratio in Gastric Cancer to Determine Recurrence Rate After Curative Resection
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/633
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Gastric Cancer
Keywords: Lymph node metastasis, Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
D2 gastrectomy is standard treatment of early gastric cancer in Japan but in other countries there is still some discord, especially in Europe and North America. Although the quantity of metastasis cancer in lymph node defines survival regardless of which country the patient is treated, the total number of lymph nodes harvested is an important factor to predict accurate staging and/or D2 gastrectomy. Both of the number total lymph nodes and the metastasis lymph node status in gastric cancer are important factors to decide each prognosis. This study evaluated the correlation between total lymph nodes retrieved and metastasis node by lymph node ratio (LNR) status to determine the recurrence rate after curative resection of gastric

DETAILED DESCRIPTION:
A retrospective chart review was made of all patients who presented with gastric cancer after curative surgery resection from January 1, 1995 to December 31, 2016 in Ramathibodi Hospital.Data of metastasis node by lymph node ratio (LNR) were evaluated. The total of lymph node less than 15 and more than 15 were evaluated. The Kaplan-Meier curve estimates recurrence survival (Log-rank test). The p-value < 0.05 is statistically significant.

OBJECTIVE :

The outcome of this study was evaluated lymph node ratio (LNR) status that determined by the ratio of total lymph node metastasis and the total lymph node which retrieved after performed the curative surgery and lymphadenectomy of gastric cancer. The correlation of LNR and prognosis of recurrence and survival of gastric cancer patients were evaluated and reported in this study.

ELIGIBILITY:
Inclusion Criteria:

* Gastric cancer after curative surgery resection
* No received neoadjuvant therapy
* Patients have tissues confirmed by Pathology
* Staging used esophagogastroduodenoscopy (EGD) or imaging, including ultrasonography, Computer Tomography (CT) or Magnetic Resonance Imaging (MRI
* Surgery was performed for curative intent and D2 lymphadenectomy and according from Japanese guideline for gastric cancer

Exclusion Criteria:

* Distant metastasis during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who presented with gastric cancer after curative surgery resection from January 1, 1995 to December 31, 2016 in Ramathibodi Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
The correlation of lymph node ratio and survival of gastric cancer patients | 5 year
  correlation of lymph node ratio and survival of gastric cancer patients.lymph node ratio was divided in to 5 ranges including 0.000-0.109, 0.110-0.209, 0.210-0.309, 0.410-0.609 and 0.610-1.000.
The correlation of lymph node ratio and prognosis of recurrence of gastric cancer patients | 5 year
  correlation of lymph node ratio and recurrence of gastric cancer patients.lymph node ratio was divided in to 5 ranges including 0.000-0.109, 0.110-0.209, 0.210-0.309, 0.410-0.609 and 0.610-1.000.

SECONDARY OUTCOMES:
The correlation of total of lymph node retrieved less than 15 and more than 15 nodes and survival of gastric cancer patients | 5 year
  correlation of total of lymph node retrieved less than 15 and more than 15 nodes and survival of gastric cancer patients..lymph node ratio was divided in to 5 ranges including 0.000-0.109, 0.110-0.209, 0.210-0.309, 0.410-0.609 and 0.610-1.000.

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Supsamutchai, MD, Study Chair — Ramathibodi Hospital
Locations (1):
- Chairat Supsamutchai, Bangkok, Bankok, Thailand

IPD SHARING:
Plan to Share IPD: No